CLINICAL TRIAL: NCT03127514
Title: Evaluation of the Safety, Tolerability, Efficacy and Activity of AMX0035, a Fixed Combination of Phenylbutyrate (PB) and Tauroursodeoxycholic Acid (TUDCA), for the Treatment of ALS
Brief Title: AMX0035 in Patients With Amyotrophic Lateral Sclerosis (ALS)
Acronym: CENTAUR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amylyx Pharmaceuticals Inc. (Industry)
Collaborators: ALS Finding a Cure (Other); ALS Association (Other); Northeast ALS Consortium (Other); Neurological Clinical Research Institute at Massachusetts General Hospital (Other); Leandro P. Rizzuto Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMX-3500
Record Dates: First submitted 2017-04-12; First posted 2017-04-25 (Actual); Results first posted 2021-08-11 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Neuromuscular Diseases; Neurodegenerative Diseases; Spinal Cord Diseases; TDP-43 Proteinopathies; Nervous System Diseases; Central Nervous System Diseases
Keywords: Randomized; Double-blind; Placebo-controlled; Amyotrophic Lateral Sclerosis; Sodium Phenylbutyrate; Tauroursodeoxycholic Acid
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Neuromuscular Diseases; Neurodegenerative Diseases; Spinal Cord Diseases; TDP-43 Proteinopathies; Nervous System Diseases; Central Nervous System Diseases | interventions — sodium phenylbutyrate and taurursodiol; 4-phenylbutyric acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo administered by mouth or via feeding tube for 24 weeks: once daily for first 3 weeks and then twice daily for remainder of study if participant tolerating
  Interventions: Other: Placebo
- AMX0035 (Experimental): AMX0035 administered by mouth or via feeding tube for 24 weeks: once daily for first 3 weeks and then twice daily for remainder of study if participant tolerating
  Interventions: Drug: AMX0035

INTERVENTIONS:
Drug: AMX0035 — AMX0035
  Other Names: Proprietary formulation of taurursodiol and sodium phenylbutyrate
  Arms: AMX0035
Other: Placebo — Matching Placebo Comparator
  Arms: Placebo

SUMMARY:
The CENTAUR trial was a 2:1 (active:placebo) randomized, double-blind, placebo-controlled Phase II trial to evaluate the safety and efficacy of AMX0035 for the treatment of ALS.

DETAILED DESCRIPTION:
AMX0035 is a combination therapy designed to reduce neuronal death through blockade of key cellular death pathways originating in the mitochondria and endoplasmic reticulum (ER). This clinical trial is designed to demonstrate that treatment is safe, tolerable, and able to slow decline in function as measured by the ALSFRS-R. The trial will also assess the effects of AMX0035 on muscle strength, vital capacity, and biomarkers of ALS including markers of neuronal death and neuroinflammation.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female, aged 18-80 years of age
2. Sporadic or familial ALS diagnosed as definite as defined by the World Federation of Neurology revised El Escorial criteria
3. Less than or equal to 18 months since ALS symptom onset
4. Capable of providing informed consent and following trial procedures
5. Slow Vital Capacity (SVC) >60% of predicted value for gender, height, and age at the Screening Visit
6. Subjects must either not take riluzole or be on a stable dose of riluzole for at least 30 days prior to the Screening Visit. Riluzole-naïve subjects are permitted in the study.
7. Women of child bearing potential (e.g. not post-menopausal for at least one year or surgically sterile) must agree to use adequate birth control for the duration of the study and 3 months after last dose of study drug. Women must not be planning to become pregnant for the duration of the study and 3 months after last dose of study drug
8. Men must agree to practice contraception for the duration of the study and 3 months after last dose of study drug. Men must not plan to father a child or provide for sperm donation for the duration of the study and 3 months after last dose of study drug

Key Exclusion Criteria:

1. Presence of tracheostomy
2. Exposure to PB, Taurursodiol or UDCA within 3 months prior to the Screening Visit or planning to use these medications during the course of the study
3. History of known allergy to PB or bile salts
4. Abnormal liver function defined as aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 3 times the upper limit of the normal
5. Renal insufficiency as defined by a serum creatinine > 1.5 times the upper limit of normal
6. Poorly controlled arterial hypertension (systolic blood pressure (SBP)>160mmHg or diastolic blood pressure (DBP)>100mmHg) at the Screening Visit
7. Pregnant women or women currently breastfeeding
8. History of cholecystectomy
9. Biliary disease which impedes biliary flow including active cholecystitis, primary biliary cirrhosis, sclerosing cholangitis, gallbladder cancer, gallbladder polyps, gangrene of the gallbladder, abscess of the gallbladder.
10. History of Class III/IV heart failure (per New York Heart Association - NYHA)
11. Severe pancreatic or intestinal disorders that may alter the enterohepatic circulation and absorption of TUDCA including biliary infections, pancreatitis and ileal resection
12. The presence of unstable psychiatric disease, cognitive impairment, dementia or substance abuse that would impair ability of the subject to provide informed consent, according to Site Investigator judgment
13. Clinically significant unstable medical condition (other than ALS) that would pose a risk to the subject if they were to participate in the study
14. Active participation in an ALS clinical trial evaluating a small molecule within 30 days of the Screening Visit
15. Exposure at any time to any biologic under investigation for the treatment of subjects with ALS (off-label use or investigational) including cell therapies, gene therapies, and monoclonal antibodies.
16. Implantation of Diaphragm Pacing System (DPS)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Yeramian, MD, Study Director — Amylyx Pharmaceuticals Inc.; Sabrina Paganoni, MD, Principal Investigator — Massachusetts General Hospital
Locations (25):
- United States (25):
  - Barrow Neurological Institute, Phoenix, Arizona
  - UC Irvine Medical Center, Orange, California
  - Forbes Norris MDA/ALS Research Center - California Pacific Medical Center, San Francisco, California
  - University of Florida Medical Center, Gainesville, Florida
  - Carol and Frank Morsini Center for Advanced Health Care - University of South Florida, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Ochsner Neuroscience Institute, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Washington University Medical Center, St Louis, Missouri
  - Neurology Associates P.C., Lincoln, Nebraska
  - Mount Sinai Beth Israel, New York, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - The Penn Comprehensive ALS Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Texas Neurology, P.A., Dallas, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - ALS Center at the Swedish Neuroscience Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Amylyx Pharmaceuticals, Inc., is in the process of developing a formal data sharing plan; requests for future data sharing can be sent to medinfo@amylyx.com

REFERENCES:
- [Background] Elia AE, Lalli S, Monsurro MR, Sagnelli A, Taiello AC, Reggiori B, La Bella V, Tedeschi G, Albanese A. Tauroursodeoxycholic acid in the treatment of patients with amyotrophic lateral sclerosis. Eur J Neurol. 2016 Jan;23(1):45-52. doi: 10.1111/ene.12664. Epub 2015 Feb 9. PMID 25664595
- [Background] Cudkowicz ME, Andres PL, Macdonald SA, Bedlack RS, Choudry R, Brown RH Jr, Zhang H, Schoenfeld DA, Shefner J, Matson S, Matson WR, Ferrante RJ; Northeast ALS and National VA ALS Research Consortiums. Phase 2 study of sodium phenylbutyrate in ALS. Amyotroph Lateral Scler. 2009 Apr;10(2):99-106. doi: 10.1080/17482960802320487. PMID 18688762
- [Derived] Bowser R, An J, Mehta L, Chen J, Timmons J, Cudkowicz M, Paganoni S. Effect of sodium phenylbutyrate and taurursodiol on plasma concentrations of neuroinflammatory biomarkers in amyotrophic lateral sclerosis: results from the CENTAUR trial. J Neurol Neurosurg Psychiatry. 2024 Jun 17;95(7):605-608. doi: 10.1136/jnnp-2023-332106. PMID 38050066
- [Derived] Paganoni S, Hendrix S, Dickson SP, Knowlton N, Berry JD, Elliott MA, Maiser S, Karam C, Caress JB, Owegi MA, Quick A, Wymer J, Goutman SA, Heitzman D, Heiman-Patterson TD, Jackson C, Quinn C, Rothstein JD, Kasarskis EJ, Katz J, Jenkins L, Ladha SS, Miller TM, Scelsa SN, Vu TH, Fournier C, Johnson KM, Swenson A, Goyal N, Pattee GL, Babu S, Chase M, Dagostino D, Hall M, Kittle G, Eydinov M, Ostrow J, Pothier L, Randall R, Shefner JM, Sherman AV, Tustison E, Vigneswaran P, Yu H, Cohen J, Klee J, Tanzi R, Gilbert W, Yeramian P, Cudkowicz M. Effect of sodium phenylbutyrate/taurursodiol on tracheostomy/ventilation-free survival and hospitalisation in amyotrophic lateral sclerosis: long-term results from the CENTAUR trial. J Neurol Neurosurg Psychiatry. 2022 May 16;93(8):871-5. doi: 10.1136/jnnp-2022-329024. Online ahead of print. PMID 35577511
- [Derived] Paganoni S, Macklin EA, Hendrix S, Berry JD, Elliott MA, Maiser S, Karam C, Caress JB, Owegi MA, Quick A, Wymer J, Goutman SA, Heitzman D, Heiman-Patterson T, Jackson CE, Quinn C, Rothstein JD, Kasarskis EJ, Katz J, Jenkins L, Ladha S, Miller TM, Scelsa SN, Vu TH, Fournier CN, Glass JD, Johnson KM, Swenson A, Goyal NA, Pattee GL, Andres PL, Babu S, Chase M, Dagostino D, Dickson SP, Ellison N, Hall M, Hendrix K, Kittle G, McGovern M, Ostrow J, Pothier L, Randall R, Shefner JM, Sherman AV, Tustison E, Vigneswaran P, Walker J, Yu H, Chan J, Wittes J, Cohen J, Klee J, Leslie K, Tanzi RE, Gilbert W, Yeramian PD, Schoenfeld D, Cudkowicz ME. Trial of Sodium Phenylbutyrate-Taurursodiol for Amyotrophic Lateral Sclerosis. N Engl J Med. 2020 Sep 3;383(10):919-930. doi: 10.1056/NEJMoa1916945. PMID 32877582
- See also: TUDCA in patients with ALS — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5024041/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults with sporadic or familial ALS were enrolled at 25 centers of the Northeast Amyotrophic Lateral Sclerosis Consortium (NEALS) in the United States from June 2017 through September 2019.
Period: Overall Study
Arm/Group | Placebo | AMX0035
Started | 48 | 89
Completed | 38 | 67
Not Completed | 10 | 22

BASELINE CHARACTERISTICS:
Population: Two participants in the AMX0035 group died soon after randomization and did not have a postbaseline efficacy assessment. These 2 participants were excluded from the primary efficacy analysis population (modified intention to treat (mITT) population), but were included in the safety population (intention to treat (ITT) population).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AMX0035 | Total
Number analyzed (Participants) | 48 | 87 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (7.6) | 57.6 (10.4) | 57.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 26 | 42
  Male | 32 | 61 | 93
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 46 | 82 | 128
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Time Since ALS Symptom Onset [Mean (Standard Deviation); unit: months] | 13.6 (3.6) | 13.5 (3.8) | 13.5 (3.8)
Bulbar Onset [Count of Participants; unit: Participants] | 10 | 26 | 36

OUTCOME MEASURES:

1. Primary Outcome: Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) Slope Change
Description: Change in slope of Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) over treatment duration. The ALSFRS-R consists of 12 items across 4 subdomains of function (bulbar, fine motor, gross motor, and breathing) with each item scored on a scale from 0 (total loss of function) to 4 (no loss of function). Total scores range from 0 to 48, with higher scores indicating better function.
Time Frame: 24 Weeks
Population: mITT population
Measure: Least Squares Mean (Standard Error); unit: Change in ALSFRS-R Total Score Per Month
Arm/Group | Placebo | AMX0035
Number analyzed (Participants) | 48 | 87
Change in ALSFRS-R Total Score Per Month | -1.66 (0.16) | -1.24 (0.12)
Statistical Analysis 1: Comparison: Placebo vs AMX0035; Test type: Superiority; p = 0.03, Mixed Models Analysis — A two-tailed P value of 0.05 or less was considered to indicate statistical significance; Random-slope, shared-baseline, linear mixed model was adjusted for age and prebaseline ALSFRS-R slope

2. Primary Outcome: Number of Participants With Adverse Events
Description: Comparison Between Groups of Number of Participants With Adverse Events Until Planned Completion
Time Frame: 24 Weeks
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | AMX0035
Number analyzed (Participants) | 48 | 89
Participants | 46 | 86

3. Primary Outcome: Number of Participants in Each Group Able to Remain on Study Drug Until Planned Discontinuation
Description: A comparison of the number of participants in each group able to remain on study drug until planned discontinuation between groups
Time Frame: 24 weeks
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | AMX0035
Number analyzed (Participants) | 48 | 87
Participants | 38 | 61

4. Secondary Outcome: Accurate Testing of Limb Isometric Strength (ATLIS) Total Score Change
Description: The ATLIS device assess the isometric muscle strength of six upper-limb and six lower-limb muscle groups. At least two trials are performed for each muscle group to assess change in rate of decline of isometric muscle strength over treatment duration. Values are standardized to the percentage of predicted normal strength based on sex, age, weight, and height. Results are presented as percent of predicted normal.
Time Frame: 24 Weeks
Population: mITT population (1 participant in the placebo group and 3 in the AMX0035 group did not have complete muscle strength data and are not included in this analysis population)
Measure: Least Squares Mean (Standard Error); unit: % of Predicted Normal Change Per Month
Arm/Group | Placebo | AMX0035
Number analyzed (Participants) | 47 | 84
% of Predicted Normal Change Per Month | -3.54 (0.26) | -3.03 (0.19)

5. Secondary Outcome: Change in Plasma Levels of Phosphorylated Axonal Neurofilament H Subunit (pNF-H)
Description: Neuronal degeneration releases phosphorylated axonal neurofilament H subunit (pNF-H) into the cerebrospinal fluid and subsequently the blood and is thought to be a potential biomarker of motor neuron degeneration; elevated plasma levels of pNF-H are presumed to correlate with neuronal injury. Change in levels of plasma pNF-H were measured from baseline to week 24
Time Frame: 24 Weeks
Population: mITT population (1 participant in the placebo group and 3 in the AMX0035 group did not have sample analyzed and are not included in this analysis population)
Measure: Least Squares Mean (Standard Error); unit: pg/ml Per Month
Arm/Group | Placebo | AMX0035
Number analyzed (Participants) | 47 | 84
pg/ml Per Month | -2.34 (4.19) | 3.58 (3.19)

6. Secondary Outcome: Rate of Decline in Slow Vital Capacity (SVC)
Description: Respiratory muscle function was assessed according to slow vital capacity (SVC). SVC was measured in an upright position for at least three trials per assessment. SVC volumes were standardized to the percentage of predicted normal value based on age, sex, and height.
Time Frame: 24 Weeks
Population: mITT population
Measure: Least Squares Mean (Standard Error); unit: % of Predicted Normal Change Per Month
Arm/Group | Placebo | AMX0035
Number analyzed (Participants) | 48 | 87
% of Predicted Normal Change Per Month | -4.03 (0.42) | -3.10 (0.31)

7. Secondary Outcome: Death, Tracheostomy, and Hospitalization
Description: The composite outcome was defined as death, a death-equivalent event (which consisted of only tracheostomy in one participant in this trial), or hospitalization, whichever occurred first; there were no instances of permanent ventilation delivered by noninvasive means in the study.
Time Frame: 24 Weeks
Population: mITT population
Measure: Number; unit: events
Arm/Group | Placebo | AMX0035
Number analyzed (Participants) | 48 | 87
events | 17 | 18

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the entire 24 week study
Description: Symptoms of ALS progression, including those consistent with disease progression were recorded as adverse events. Any worsening of a disease progression measure that was being analyzed separately (ALSFRS-R, ATLIS, and SVC) was not recorded as an adverse event
Arm/Group | Placebo | AMX0035
All-Cause Mortality (participants affected / at risk) | 2/48 | 5/89
Serious Adverse Events (participants affected / at risk) | 9/48 | 11/89
Other Adverse Events (participants affected / at risk) | 46/48 | 86/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=48) | AMX0035 (N=89)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 1
Catheter Site Infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Device dislocation (Product Issues) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=48) | AMX0035 (N=89)
Diarrhoea (Gastrointestinal disorders) | 8 | 19
Constipation (Gastrointestinal disorders) | 12 | 12
Nausea (Gastrointestinal disorders) | 6 | 16
Abdominal pain (Gastrointestinal disorders) | 4 | 7
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 10
Dry mouth (Gastrointestinal disorders) | 4 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 4
Abdominal discomfort (Gastrointestinal disorders) | 0 | 5
Dysphagia (Gastrointestinal disorders) | 4 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Fall (Injury, poisoning and procedural complications) | 18 | 25
Contusion (Injury, poisoning and procedural complications) | 4 | 5
Laceration (Injury, poisoning and procedural complications) | 3 | 6
Headache (Nervous system disorders) | 11 | 13
Dizziness (Nervous system disorders) | 2 | 9
Viral Upper Respiratory Tract Infection (Infections and infestations) | 2 | 10
Urinary Tract Infection (Infections and infestations) | 3 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Alanine aminotransferase increased (Investigations) | 3 | 4
Aspartate aminotransferase increased (Investigations) | 3 | 4
Weight decreased (Investigations) | 1 | 5
Fatigue (General disorders) | 3 | 7
Oedema peripheral (General disorders) | 3 | 2
Asthenia (General disorders) | 0 | 5
Rash (Skin and subcutaneous tissue disorders) | 4 | 5
Insomnia (Psychiatric disorders) | 3 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/14/NCT03127514/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/14/NCT03127514/SAP_001.pdf